CLINICAL TRIAL: NCT06525727
Title: External Validation of the Falls Decision Rule to Exclude Intracranial Bleeding Without Head CT in Geriatric Patients Presenting to the Emergency Department With A Fall
Brief Title: Validation of Falls Decision Rule to Exclude Intracranial Bleeding in Geriatric Fall Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Sinan Karacabey, Assoc. Prof., Marmara University
Other Study IDs: 12.01.2024.48
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Hemorrhages
Keywords: Falls Rule; geriatric; rule; external validation
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 65 years and over: Patients aged 65 years and over who came to the emergency department with a fall on level ground ((either inside or outside), off a chair, toilet seat or out of bed) within the last 48 hours
  Interventions: Other: Falls Decision Rule

INTERVENTIONS:
Other: Falls Decision Rule — The Falls Decision Rule is a rule used to assess the risk of intracranial haemorrhage in geriatric patients and to prevent brain tomography (CT) in low-risk patients. This rule recommends that brain CT is not necessary in patients who do not have significant head trauma, memory loss, newly developing neurological examination disorder, or frailty score lower than 5 after a fall.

SUMMARY:
Although falls are the most important cause of intracranial hemorrhage in the population over 65, studies have shown that bleeding occurs in only 5% of geriatric patients who fall. Guidelines have been developed to assist the clinician in identifying patients at risk of intracranial hemorrhage due to the relatively low incidence but significant morbidity and mortality. The 'Falls Decision Rule' was developed by de Wit et al. in 2023 to assess the need for CT in this patient group. In this study, external validation of this newly developed score was planned to evaluate its safety, applicability, and authenticity.

DETAILED DESCRIPTION:
In the geriatric population (≥65 years), falls are responsible for 70% of traumatic brain injury. Computed tomography (CT) evaluation of the brain used in evaluating these patients makes it possible to detect intracranial hemorrhage in the early period. Thus, it plays a critical role in initiating timely and necessary interventions. These interventions include blood pressure control, hemorrhage control, and neurosurgical interventions.

Although the most important cause of intracranial hemorrhage in this population is falls, studies have shown that bleeding occurs in only 5% of geriatric patients who fall. Therefore, it is inefficient and costly to perform brain CT evaluation in every patient.

Rules have been developed to assist the clinician in identifying patients at risk of intracranial hemorrhage, which has a relatively low incidence but significant morbidity and mortality. The Canadian Brain CT rule, one of the most widely used rules for this purpose, determines the need for brain CT in patients with head trauma. However, this rule applies to patients with disorientation, amnesia, or loss of consciousness. There are insufficient studies to guide neuroimaging for older adults who hit their heads while falling but do not experience these symptoms. In addition, guidance from the literature for older adults who fall but cannot describe what happened or did not hit their heads is also insufficient. The 'Falls Decision Rule' was developed by de Wit et al. in 2023 to assess the need for CT in this patient group. This criterion was developed by including a total of 4308 patients in the United States and Canadian emergency departments. It suggests that in patients in the geriatric population, there is no need for Brain CT in the absence of significant head trauma due to falls, no memory loss due to falls, no newly developing neurological examination disorder, and a clinical frailty score of less than 5. The sensitivity of this score to exclude clinically significant bleeding is 98.6% (95% CI 94.9-99.6), and the negative predictive value is 99.8% (95% CI 99.2-99.8).

This newly developed rule was developed only in a specific geographical region. In this study, external validation of this newly developed score was planned in order to evaluate its safety, applicability, and accuracy.

Patients over 65 years of age who come to the emergency department with a fall will be observationally recorded on the case form after obtaining consent from the patient or his/her relatives and will be followed up for clinically significant intracranial hemorrhage within 42 days. This study is a validation study, and the protocol used in the original study will be followed. The study is a prospective observational study. The study will start after ethics committee approval and will be conducted at Marmara University Pendik Training and Research Hospital. The data collection process will be completed when the targeted sample size is reached.

The sample size was calculated for the diagnostic value study planned to validate the fall decision rule developed by de Wit et al. to rule out patients with intracranial hemorrhage. Using the incidence, sensitivity, and specificity values shared by the authors as a reference, the minimum sample size to be included in the study was calculated as 663, with 80% power and 0.05% margin of error. Considering the risk of missing and inaccurate measurements, the target sample size was increased by 15% and set as 763.

Data will be obtained from patient files, Hospital Information Management System, and PACS systems; Demographic information (age, gender), Known diseases (HT, DM, AF, CHF, etc.), Information on falls, Physical examination information), Consultation notes, if any, Antiplatelet, anticoagulant use, Frailty score, The CT scan results will be saved.

Patients will be followed up for delayed intracranial hemorrhage within 42 days after the fall as in the original study. Also as in the methodology of the original study, patients will be followed up through the electronic information system. Previous studies have shown that this method has a low sensitivity (37%, 95% CI 21-56) for intracranial hemorrhage when patients are questioned for intracranial hemorrhage by telephone call. Therefore, in the original study and this study, it was planned to follow up the information of the patients from the electronic information system records instead of telephoning. The intracranial hemorrhage status of the patients within 42 days will be followed up through the hospital information system and patient information system.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older.
* Patients who presented to the emergency department within 48 hours of a fall.
* Patients who provided informed consent to participate in the study or whose legal guardians provided consent if the patients are unable to do so.

Exclusion Criteria:

* Patients who have already been included in the study previously.
* Patients who refuse medical treatment or withdraw consent during the study period.
* Patients with incomplete data necessary for the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of geriatric patients aged 65 years and older who present to the emergency department within 48 hours of experiencing a fall on level ground ((either inside or outside), off a chair, toilet seat, or out of bed). These patients will be included if they provide informed consent or if their legal guardians provide consent if the patients are unable to do so. The study aims to externally validate the Falls Decision Rule to exclude intracranial bleeding in this specific population. All patients meeting the inclusion criteria and none of the exclusion criteria will be enrolled in the study, and they will be observed for clinically significant intracranial bleeding for up to 42 days post-fall.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gray I, de Wit K. Fast-tracking falls - expediting emergency care with evidence. CJEM. 2025 Aug;27(8):580-581. doi: 10.1007/s43678-025-00970-x. No abstract available. PMID 40856903
- [Result] Kudu E, Altun M, Danis F, Karacabey S, Sanri E, Denizbasi A. Validating the falls decision rule: optimizing head CT use in older adults with ground-level falls. CJEM. 2025 Aug;27(8):629-637. doi: 10.1007/s43678-025-00937-y. Epub 2025 May 13. PMID 40360963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited patients aged 65 years and older who presented to the emergency department of Marmara University Pendik Training and Research Hospital within 48 hours of a fall on level ground, from a chair, toilet seat, or out of bed. Recruitment began on January 20, 2024, and continued until the required sample size was reached on October 1, 2024, ensuring adequate participant inclusion.
Groups:
- Patients Who Did Not Undergo Head CT Scan on Index Visit: This group includes patients aged 65 years and older who presented to the emergency department following a ground-level fall but did not undergo head CT imaging during their initial visit. The decision not to perform a CT scan was made by the treating emergency physician based on clinical assessment and existing decision rules. These patients were monitored for delayed intracranial bleeding through a 42-day follow-up period.
- Patients Who Underwent Head CT Scan on Index Visit: This group includes patients aged 65 years and older who presented to the emergency department following a ground-level fall and underwent head CT imaging during their initial visit. The decision to perform a CT scan was made by the treating emergency physician based on clinical assessment and existing decision rules. These patients were evaluated for intracranial bleeding at the time of presentation and monitored for delayed bleeding through a 42-day follow-up period.
Period: Overall Study
Arm/Group | Patients Who Did Not Undergo Head CT Scan on Index Visit | Patients Who Underwent Head CT Scan on Index Visit
Started | 259 | 541
Completed | 259 | 541
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Identified With CIIB on Initial Visit and 42 Day Follow-up: This group includes patients aged 65 years and older who were diagnosed with clinically important intracranial bleeding (CIIB) either at the initial emergency department visit or during the 42-day follow-up period. CIIB was defined as intracranial bleeding requiring medical or surgical intervention or resulting in mortality. Patients in this group were managed according to clinical guidelines, and those not initially identified with CIIB were closely monitored for delayed bleeding.
- Patients Without CIIB: This group includes patients aged 65 years and older who were not diagnosed with clinically important intracranial bleeding (CIIB) during the initial emergency department visit or the 42-day follow-up period. These patients either did not undergo head CT or had a negative CT result at presentation, with no subsequent evidence of intracranial bleeding requiring medical or surgical intervention. Additionally, they exhibited no signs of bleeding throughout the follow-up period and did not experience fatal outcomes related to CIIB.
- Total: Total of all reporting groups
Arm/Group | Patients Identified With CIIB on Initial Visit and 42 Day Follow-up | Patients Without CIIB | Total
Number analyzed (Participants) | 49 | 751 | 800
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 80.0 [71.5 to 88.0] | 78.0 [72.0 to 84.0] | 78.0 [72.0 to 85.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 457 | 479
  Male | 27 | 294 | 321
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 49 | 751 | 800
Confirmed history of head trauma [Count of Participants; unit: Participants] | 41 | 407 | 448
Unclear history of head trauma [Count of Participants; unit: Participants] | 3 | 36 | 39
Confirmed history of amnesia of events [Count of Participants; unit: Participants] | 20 | 69 | 89
Unclear history of amnesia of events [Count of Participants; unit: Participants] | 12 | 27 | 39
Clinical Frailty Scale score [Count of Participants; unit: Participants]
  1 Healthy, active and very fit | 3 | 85 | 88
  2 No disease symptoms, occasional exercise | 9 | 170 | 179
  3 Controlled medical issues, walk only | 11 | 210 | 221
  4 Symptoms limit activities | 5 | 113 | 118
  5 Need help with daily living activities^ | 2 | 69 | 71
  6 Need help with bathing/dressing | 9 | 53 | 62
  7-8 Completely dependent for everything | 9 | 44 | 53
  9 Terminally ill, life expectancy < 6 months | 1 | 7 | 8
Abnormal neurological examination from baseline [Count of Participants; unit: Participants] | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Clinically Important Intracranial Bleeding
Description: The primary outcome is 'clinically significant intracranial hemorrhage' identified within 42 days following the initial presentation in the emergency department. 'Clinically significant intracranial hemorrhage' is defined as hemorrhage within the cranial vault, encompassing subdural, intracerebral, intraventricular, subarachnoid, epidural hemorrhage, and cerebral contusion, necessitating medical or surgical intervention. Medical intervention is defined as any of the following actions: temporary or permanent cessation of anticoagulant or antiplatelet medications; administration of an antifibrinolytic agent; reversal of anticoagulation; or hospitalization for neurological monitoring. These criteria align with those established in the original study.
Time Frame: From baseline to 42 days (Patients will be followed up for 42 days after the fall and evaluated for delayed intracranial haemorrhage).
Measure: Count of Participants; unit: Participants
Groups:
- Patients Need Head CT According to Falls Decision Rule: Based on the Falls Decision Rule, a head CT scan is recommended for patients who meet any of the following criteria:
  * History of head trauma during the fall.
  * New abnormalities on neurological examination upon ED presentation.
  * Memory loss (amnesia) regarding the events surrounding the fall.
  * Clinical Frailty Scale score of 5 or higher.
- Patients do Not Need Head CT According to Falls Decision Rule: Based on the Falls Decision Rule, patients who do not require a head CT scan must meet all of the following criteria:
  * No history of head trauma during the fall.
  * No new abnormalities on neurological examination.
  * No memory loss (amnesia) regarding the events surrounding the fall.
  * A Clinical Frailty Scale score of less than 5.
Arm/Group | Patients Need Head CT According to Falls Decision Rule | Patients do Not Need Head CT According to Falls Decision Rule
Number analyzed (Participants) | 559 | 241
Participants | 48 | 1
Statistical Analysis 1: Comparison: Patients Need Head CT According to Falls Decision Rule vs Patients do Not Need Head CT According to Falls Decision Rule; The primary objective of the study was to assess the external validation of the Falls Decision Rule. In this evaluation, patients were categorized into two groups based on the rule: those for whom a CT scan was recommended and those for whom it was not; Test type: Other; Diagnostic accuracy; Diagnostic performance was analyzed in terms of sensitivity, specificity, NPV, PPV and likelihood ratios, all reported with 95% confidence interval; Sensitivity = 97.96, 95% CI 2-sided [89.15 to 99.95]
Statistical Analysis 2: Comparison: Patients Need Head CT According to Falls Decision Rule vs Patients do Not Need Head CT According to Falls Decision Rule; Test type: Other; Diagnostic accuracy; Specificity = 31.96, 95% CI 2-sided [28.63 to 35.42]
Statistical Analysis 3: Comparison: Patients Need Head CT According to Falls Decision Rule vs Patients do Not Need Head CT According to Falls Decision Rule; Test type: Other; Diagnostic accuracy; Negative predictive value = 99.59, 95% CI 2-sided [97.17 to 99.94]
Statistical Analysis 4: Comparison: Patients Need Head CT According to Falls Decision Rule vs Patients do Not Need Head CT According to Falls Decision Rule; Test type: Other; Diagnostic accuracy; Positive predictive value = 8.59, 95% CI 2-sided [8.1 to 9.1]
Statistical Analysis 5: Comparison: Patients Need Head CT According to Falls Decision Rule vs Patients do Not Need Head CT According to Falls Decision Rule; Test type: Other; Diagnostic accuracy; Negative likelihood ratio = 0.06, 95% CI 2-sided [0.01 to 0.42]
Statistical Analysis 6: Comparison: Patients Need Head CT According to Falls Decision Rule vs Patients do Not Need Head CT According to Falls Decision Rule; Test type: Other; Diagnostic accuracy; Positive likelihood ratio = 1.44, 95% CI 2-sided [1.35 to 1.53]

2. Secondary Outcome: Number of Participant With Neurosurgical Intervention
Description: Neurosurgical intervention was defined as any surgical procedure performed to manage clinically important intracranial bleeding (CIIB) identified either at the initial emergency department visit or during the 42-day follow-up period.
Time Frame: 42 day
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Identified With CIIB on Initial Visit and 42 Day Follow-up | Patients Without CIIB
Number analyzed (Participants) | 49 | 751
Participants | 6 | 0

3. Secondary Outcome: Number of Patients With Mortality
Description: Mortality was defined as death occurring at any point during the 42-day follow-up period, regardless of whether it was directly attributed to clinically important intracranial bleeding (CIIB). Deaths were identified through national healthcare system.
Time Frame: 42 day
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Identified With CIIB on Initial Visit and 42 Day Follow-up | Patients Without CIIB
Number analyzed (Participants) | 49 | 751
Participants | 12 | 34

ADVERSE EVENTS:
Time Frame: Deaths assessed through 42 days
Description: Since this is an observational study, no direct interventions or experimental treatments were applied to the participants. Therefore, the likelihood of observing adverse events directly related to the study itself is nonexistent. Only all-cause mortality was assessed through 42 days.
Arm/Group | Patients Identified With CIIB on Initial Visit and 42 Day Follow-up | Patients Without CIIB
All-Cause Mortality (participants affected / at risk) | 12/49 | 34/751
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study has limitations, primarily its single-center design, which may limit generalizability. However, as an external validation study, the findings suggest applicability to broader populations. Variability in physician judgment on CT use is another limitation, despite standardized training. Not all patients underwent CT at the initial visit, posing a risk of missed CIIB. However, a 42-day follow-up ensured comprehensive assessment, with no patients lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT06525727/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT06525727/SAP_001.pdf